CLINICAL TRIAL: NCT03708926
Title: Effect of Abaloparatide on Lumbar Disc Degeneration
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to obtain drugs from supplier.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00185784
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2020-05

CONDITIONS: Degeneration Disc Intervertebral
Keywords: degenerative disc disease; low back pain; PTH; abaloparatide
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain | interventions — abaloparatide; Parathyroid Hormone-Related Protein

STUDY DESIGN:
Intervention Model Description: placebo controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- abaloparatide (Experimental): abaloparatide 80 mcg subcutaneously once daily for 90 days
  Interventions: Drug: Abaloparatide
- placebo (Placebo Comparator): placebo formulated similarly but without active abaloparatide injected subcutaneously once daily for 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abaloparatide — abaloparatide injection pen
  Other Names: Tymlos, PTHrP
  Arms: abaloparatide
Drug: Placebo — placebo injection pen
  Arms: placebo

SUMMARY:
Low back pain is a major public health issue as the leading cause of disability globally. Degeneration of intervertebral disc (IVD) disorder is once source of low back pain. Current treatment options for low back pain secondary to degeneration of intervertebral disc include conservative care, steroid injections, prescription pain medications, physical therapy, or surgery, such as discectomy or laminectomy. Treatments focus on addressing manifested symptoms rather than functional causes, and symptomatic treatment of discogenic low back pain is less than ideal. The investigators have recently found that parathyroid hormone (PTH) effectively attenuates disc degeneration in aged mice. This clinical trial will test if 3-months of daily PTH-related protein (PTHrP), abaloparatide will improve pain, function, and disc health in people with low back pain secondary to lumbar disc degeneration.

DETAILED DESCRIPTION:
The investigators will perform a randomized, double blind, placebo controlled proof-of-concept Phase 2 clinical trial of the effect of abaloparatide for the treatment of lumbar degenerative disc disease. Adults with clinically significant lumbar degenerative disc disease who meet inclusion and exclusion criteria and sign informed consent with be randomized in a 2:1 ratio to study drug:placebo.

The study team physicians will review pertinent laboratory data, medication history, and problem lists in the potential research participant's medical record to ensure eligibility for the study. The investigators will also contact the potential research participants by telephone to explain the study in further detail and elicit information not available in the medical record that would affect the potential participant's eligibility to participate in the study.

Potential research participants who meet the study criteria and are interested in participating in the study will have an appointment arranged at the Johns Hopkins Orthopedic Clinic. At the study visit, a study team physician and research coordinator will review the study and consent the research participants.

Research participants who provide informed consent will have age, sex, and ethnicity recorded, undergo a focused history and physical exam, and have any necessary blood samples collected for inclusion/exclusion criteria. The focused history will include the age of onset of symptoms, age at diagnosis of degenerative disc disease, mechanism of injury, treatments utilized, and the research participant's current perception of his or her disease control. The focused physical exam will include inspection and palpation of the affected sites to assess for pain and mobility of the spine. Research participants will be asked to rate current pain attributed to degenerative disc disease on a Likert scale pain level and asked to fill out the Oswestry Disability Index (ODI) and Patient-Reported Outcomes Measurement Information System (PROMIS-29) and have spinal x-rays and an MRI of the lumbar spine obtained.

One hundred nine people who meet the study criteria and provide informed consent will be randomly assigned to 2 groups (abaloparatide:placebo) in a 2:1 fashion (n=73 abaloparatide; 36 placebo).

Participants will be taught how to self-administer a injection of the study drug. Participants and the study doctor will not know if the participant is receiving abaloparatide or placebo as the study drug. Participants will inject the study drug daily for 3 months.

Blood and urine samples will be collected 2 weeks after study initiation to evaluate clinical safety.

Physical exams, health questionnaires, and MRI scans will be performed at 3-, 6-, and 12-month follow-up visits.

The trial will be blinded for all the investigators acquiring and analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic moderate to severe discogenic low back pain as defined by centralized chronic low back pain with a discogenic character (i.e. increases with activity, worsened with sitting or standing, or requires frequent change of positions) and has been present for 6+ months
* Identifiable change in disc morphology as defined by MRI consistent with early degenerative disc disease as defined by both Modified Pfirrmann (MRI) score of 2-3 (Graded 1-8, where 1= hydrated healthy disc, 8 = dark, dehydrated disc) and Modic Grade II change or less
* Single- or two-level DDD at lumbar spine
* < 30% vertebral body height loss
* Oswestry disability index score > 30
* Failed > 3 months of appropriate non-operative care (i.e. pain medication, local drug injections, physical therapy)
* Predominant back pain with or without leg pain
* Able and willing to comply with follow-up schedule
* Willing to give written informed consent

Exclusion Criteria:

* Presence of objective motor deficit
* Symptomatic compressive pathology due to stenosis or disc herniation
* Any spondylolisthesis
* Any spondylolysis
* Scoliosis > 20 degrees
* Spinal tumor
* Previous thoracic or lumbar fusion
* Current or prior fracture at T10-S1
* Arachnoiditis
* Current or prior use of PTHrP (abaloparatide) or PTH (teriparatide) analog
* Diagnosis of osteoporosis or osteopenia that is not well controlled on anti-resorptive therapy and anticipated to require use of an anabolic agent, such as abaloparatide or teriparatide.
* Evidence of metabolic bone disease as evidenced by abnormalities in calcium, intact parathyroid hormone, phosphorus or alkaline phosphatase in blood or elevated spot urine calcium to creatinine ratio.
* History of or current osteosarcoma or cancer metastatic to the bone
* History of or current Paget's disease of bone
* History of or current nephrolithiasis
* History of or current multiple myeloma
* History of focal radiation to any bone
* Current Pregnancy or breastfeeding
* Current use of medications that increase risk of hypercalcemia, such as thiazide diuretics
* Diagnosis of psychotic disorder
* Participation in another study on investigational drug
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with improvement in symptomatic or radiographic symptoms as indicated by composite score aggregated from the Oswestry Disability Index (ODI) and Pfirrmann grading system | 6 months
  Composite score will be graded as a score of 0, 1 or 2, whereas:
  * 0 (no improvement) = less than 15 point score improvement on Oswestry Disability Index (ODI) and less than 1 grade improvement on Pfirrmann grading system.
  * 1 (some improvement - symptomatic or radiographic) = 15 point or greater improvement on ODI score OR at least 1 grade improvement on Pfirrmann grading system.
  * 2 (definite improvement) = 15 point or greater improvement on ODI score AND 1 grade or greater improvement on Pfirrmann grading system.
  ODI is scored on a scale of 0-100 with higher scores indicating worse disability. A decrease in ODI of 15 points is considered a clinically (symptomatic) meaningful improvement by the FDA. The modified Pfirrmann Grading system is an MRI based score (radiographic) of disc degeneration on a scale of 1-8, with higher scores indicating more severe degeneration, such that improvement is by decreasing score.

SECONDARY OUTCOMES:
Change in disability as assessed by ODI | Baseline, 3 months, 6 months, 12 months
  The efficacy of abaloparatide on disability will be assessed by absolute difference in ODI from baseline in abaloparatide versus placebo group, reported as average per group. ODI assessed pain related disability is scored on a scale of 0-100 with higher scores indicating worse disability.
Change in clinically significant improvement in disability as assessed by ODI | Baseline, 3 months, 6 months, 12 months
  The efficacy of abaloparatide on disability will be assessed by percentage of patients with 15 point or greater improvement in ODI from baseline in abaloparatide versus placebo group. ODI assessed pain related disability is scored on a scale of 0-100 with higher scores indicating worse disability. A decrease in ODI of 15 points is considered a clinically meaningful improvement by the FDA.
Change in pain as assessed by pain numerical rating scale | Baseline, 3 months, 6 months, 12 months
  The efficacy of abaloparatide on disability will be assessed by absolute difference in pain numerical rating scale from baseline in abaloparatide versus placebo group, reported as average per group. The pain numerical rating scale assesses pain intensity on a scale of 0-10 with higher scores indicating worse pain.
Change in disability as assessed by PROMIS-29 score | Baseline, 3 months, 6 months, 12 months
  The efficacy of abaloparatide on disability will be assessed by absolute change in PROMIS-29 score from baseline in abaloparatide versus placebo group, reported as average per group. The PROMIS-29 is a multi-dimensional quality of life instrument that assesses pain, physical function, fatigue, anxiety, depression, sleep disturbance, and social participation on a scale of 0-100 with higher scores indicating more disturbances of that dimension.
Change in radiographic markers of Degenerative Disc Disease (DDD) as assessed by absolute difference in Pfirrmann Grading system | Baseline, 3 months, 6 months, 12 months
  The efficacy of abaloparatide on changes in radiographic markers of DDD will be assessed by absolute difference in modified Pfirrmann Grading system from baseline, reported as average per group. The modified Pfirrmann Grading system is an MRI based score of disc degeneration on a scale of 1-8, with higher scores indicating more severe degeneration.
Change in radiographic markers of DDD as assessed by improvement in Pfirrmann Grading system | Baseline, 3 months, 6 months, 12 months
  The efficacy of abaloparatide on radiographic markers of DDD will be evaluated using the percentage of patients with 1 grade or greater improvement in modified Pfirrmann Grading system from baseline in the abaloparatide versus placebo group. The modified Pfirrmann Grading system is an MRI based score of disc degeneration on a scale of 1-8, with higher scores indicating more severe degeneration.
Change in radiographic markers of DDD as assessed by average absolute difference in Modic score | Baseline, 3 months, 6 months, 12 months
  The efficacy of abaloparatide on radiographic markers of DDD will be assessed by absolute difference in Modic Score from baseline, reported as average per group. Modic score is an MRI based score characterizing the vertebral endplate. Modic score correlates with progressive degenerative changes in the endplate, where 0 = normal; 1= hypervascular; 2 = fatty infiltration; 3 = sclerosis.
Change in radiographic markers of DDD as assessed by Modic score | Baseline, 3 months, 6 months, 12 months
  The efficacy of abaloparatide on radiographic markers of DDD will be evaluated using percentage of patients with 1 grade or greater improvement in Modic Score from baseline in the abaloparatide versus placebo group. Modic score is an MRI based score characterizing the vertebral endplate. Modic score correlates with progressive degenerative changes in the endplate, where 0 = normal; 1= hypervascular; 2 = fatty infiltration; 3 = sclerosis.
Change in pain management based on analgesic usage | Baseline, 3 months, 6 months, 12 months
  Evaluate change in pain management in abaloparatide versus placebo groups based on change in the dosage of analgesic used and the number of days of back pain (longer than 30 min/day) in week prior to baseline compared to week prior to 3-, 6-, and 12-month visits.
Requirement of surgical intervention for back pain by patients | 12 months
  Proportion of patients proceeding to a surgical intervention within the 12-month study period in the abaloparatide versus placebo group will be assessed by percentages per arm
Requirement of escalation of medical care related to back pain by patients | 12 months
  Proportion of patients requiring escalation of medical care related to back pain (e.g. spine surgery, injections into IVD, or Emergency Department visits related to debilitating back pain) will be assessed by percentages per arm

CONTACTS AND LOCATIONS:
Overall Officials: Janet Crane, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No